CLINICAL TRIAL: NCT05151055
Title: A Randomized, Double-Blind, Placebo-Controlled Trial To Determine The Safety and Efficacy of Lactoferrin With Vitamin E and Zinc as an Oral Therapy for Mild to Moderate Hormonal Acne in Adult Women
Brief Title: Lactoferrin + Vitamin E + Zinc for Hormonal Acne
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: United Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD2019-01
Record Dates: First submitted 2021-11-28; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Hormonal Acne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactezin (Experimental): 100 mg lactoferrin, 11 IU vitamin E (as alpha tocopherol), and 5 mg zinc (as zinc gluconate)
  Interventions: Dietary Supplement: Lactezin
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactezin — 100 mg lactoferrin, 11 IU vitamin E (as alpha tocopherol), and 5 mg zinc (as zinc gluconate)
  Arms: Lactezin
Dietary Supplement: Placebo — starch
  Arms: Placebo

SUMMARY:
We previously showed that twice daily intake of a combination of 100 mg lactoferrin, 11 IU vitamin E, and 5 mg zinc significantly reduced both inflammatory and non-inflammatory acne lesions compared to placebo control. In that study, females showed an overall better response compared to males in terms of total lesions. We speculated that the gender effect may be due to mitigation of the pre- menstrual flare-ups women have that lead to recurring acne, making them have a better response. The objectives of this study are: 1.) to characterize the efficacy and safety of 100 mg lactoferrin + 11 IU vitamin E + 5 mg zinc in the adult female population who suffer from hormonal acne, 2.) to determine whether the anti-acne effect is maintained after treatment stops.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 22-50.
2. At least 3 inflammatory acne lesions, mostly found on (but not limited to) the lower face
3. Not responsive to conventional treatment
4. Clinical diagnosis of mild to moderate acne according to Lehmann et. al.

Exclusion Criteria:

1. Females who are pregnant (confirmed by a pregnancy test), breast- feeding, or planning a pregnancy.
2. Post-menopausal women
3. Current or recent (within 3 months) use of any topical or oral anti- acne products,
4. Hormonal contraceptive intake in the preceding six months
5. A cancer diagnosis within the past 5 years
6. History of hypersensitivity to any component of the test product.
7. Current imuunosuppression. Specifically, these include patients with co-morbidities such as diabetes, HIV, chronic diseases patients requiring maintenance medications, such as vascular disease,

   * hepatitis, eczema, psoriasis, or acute febrile/infectious illnesses
   * (i.e. Dengue, pneumonia, etc)

Ages: 22 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Mean percentage change in inflammatory acne lesions at 2, 4, 6, 8, 10, and 12 weeks compared to baseline, in the treatment versus placebo groups | 12 weeks

SECONDARY OUTCOMES:
Percentage change in inflammatory acne lesion counts at 14, 16, 18, 20, 22, and 24 weeks compared to baseline | 24 weeks
Mean percent change in the AFAST scores at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 weeks compared to baseline, in the treatment versus placebo groups | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Management and Testing Associates, Inc., City of Muntinlupa, Philippines

IPD SHARING:
Plan to Share IPD: No